CLINICAL TRIAL: NCT00892554
Title: The Impact of Docosahexaenoic Acid on Neuropsychological Status in Females With Phenylketonuria
Brief Title: The Effect of Supplemental Docosahexaenoic Acid (DHA) on Neurocognitive Outcomes in Teen and Adult Women With Phenylketonuria(PKU)
Acronym: PKU&DHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Atlanta Clinical and Translational Science Institute (Other)
Responsible Party: Principal Investigator, Rani Singh, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00002447
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Phenylketonuria
Keywords: Phenylketonurias; Docosahexaenoic Acids; Neuropsychological Tests; Female; Adolescent; Adult
MeSH Terms: conditions — Phenylketonurias | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA supplementation (Experimental)
  Interventions: Dietary Supplement: Docosahexaenoic Acid
- corn/soy capsule, no DHA (Placebo Comparator)
  Interventions: Dietary Supplement: Corn/soy oil

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic Acid — Capsules providing 10 mg DHA/kg body weight/day taken once daily
  Other Names: DHASCO-S
  Arms: DHA supplementation
Dietary Supplement: Corn/soy oil — Capsules taken once daily
  Arms: corn/soy capsule, no DHA

SUMMARY:
The purpose of this study is to determine if taking supplemental DHA improves measures of processing speed and executive function in teen and adult women with PKU.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Phenylketonuria
* Ages 12 years and older
* Able to complete neuropsychological testing

Exclusion Criteria:

* Pregnancy
* Currently taking DHA supplement

Ages: 12 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Cognitive processing speed | 0 months, 4.5 months
Executive function | 0 months, 4.5 months

SECONDARY OUTCOMES:
Plasma and red blood cell DHA concentrations | 0 months, 4.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Rani H. Singh, PhD, RD, LD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Yi SH, Kable JA, Evatt ML, Singh RH. A randomized, placebo-controlled, double-blind trial of supplemental docosahexaenoic acid on cognitive processing speed and executive function in females of reproductive age with phenylketonuria: A pilot study. Prostaglandins Leukot Essent Fatty Acids. 2011 Dec;85(6):317-27. doi: 10.1016/j.plefa.2011.09.004. Epub 2011 Oct 14. PMID 22000478
- See also: PKU & DHA Study Website — http://genetics.emory.edu/NUTRITION/pku_dha_study/